CLINICAL TRIAL: NCT02354105
Title: A Noninterventional Study to Assess the Effectiveness of Certolizumab Pegol in Patients With Axial Spondyloarthritis in Daily Practice
Brief Title: A Study to Assess the Effectiveness of Certolizumab Pegol in Patients With Axial Spondyloarthritis in Daily Life
Acronym: CIMAX
Status: Completed | Type: Observational
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: AS0002
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial Spondyloarthritis; Radiographic Axial Spondyloarthritis; Non-radiographic Axial Spondyloarthritis; Ankylosing spondylitis; Diagnosis; Cimzia; CZP; Certolizumab Pegol; CDP870
MeSH Terms: conditions — Axial Spondyloarthritis; Non-Radiographic Axial Spondyloarthritis; Spondylitis, Ankylosing; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CZP treatment: axSpA patients who have been newly prescribed Certolizumab Pegol (CZP).

SUMMARY:
The primary purpose is to assess the effectiveness of certolizumab pegol in patients with axial spondyloarthritis under routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* The patient personally signed and dated a Patient Data Consent Form (PDCF) prior to Visit 2. No data can be entered into the electronic Documentation form (eDF) prior to signature of the PDCF.
* The patient must have a clinical diagnosis of active axial spondyloarthritis (axSpA), [ankylosing spondylitis (AS) or nonradiographic axial spondyloarthritis (nr-axSpA)] according to the diagnostic criteria used by the physician in routine clinical practice.
* The decision to prescribe Certolizumab Pegol (CZP) is made by the physician independent of the patient's participation in the NIS.
* The patient must be newly prescribed CZP according to local regulations or guidelines (eg, Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) >=4).
* Treatment is according to instructions in the Summary of Product Characteristics (SmPC) for patients considered by the treating physician to be reliable and capable of adhering to the observational plan (eg, able to understand and complete questionnaires).
* If a patient is participating in an ongoing investigational study, then he/she will not be able to take part in this study.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with axial spondyloarthritis (axSpA) (including both ankylosing spondylitis (AS) and nonradiographic axial spondyloarthritis (nr-axSpA)) who have been newly prescribed Certolizumab Pegol (CZP) by the treating physician in regular course of practice.
Sampling Method: Non-Probability Sample
Enrollment: 680 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 52 in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in the overall axial spondyloarthritis (axSpA) population, and the ankylosing spondylitis (AS) and nonradiographic axSpA (nr-axSpA) subpopulations | From Baseline to Week 52
  The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in the overall axSpA population, and the AS and nr-axSpA subpopulations | From Baseline to Week 12
  The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.
Change from Baseline to Week 24 in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in the overall axSpA population, and the AS and nr-axSpA subpopulations | From Baseline to Week 24
  The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 to 10, with lower scores indicating lower disease activity.
Assessment of SpondyloArthritis International Society 20 % (ASAS20) response criteria in the overall axSpA population, and the AS and nr-axSpA subpopulations at Week 12 | At Week 12
  The ASAS20 response is the improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PtGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain.
Assessment of SpondyloArthritis International Society 20 % (ASAS20) response criteria in the overall axSpA population, and the AS and nr-axSpA subpopulations at Week 24 | At Week 24
  The ASAS20 response is the improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PtGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain.
Assessment of SpondyloArthritis International Society 20 % (ASAS20) response criteria in the overall axSpA population, and the AS and nr-axSpA subpopulations at Week 52 | At Week 52
  The ASAS20 response is the improvement of at least 20 % and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PtGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and absence of deterioration in the potential remaining domain.
Assessment of SpondyloArthritis International Society 40 % (ASAS40) response criteria in the overall axSpA population, and the AS and nr-axSpA subpopulations at Week 12 | At Week 12
  The ASAS40 response is the relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PtGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
Assessment of SpondyloArthritis International Society 40 % (ASAS40) response criteria in the overall axSpA population, and the AS and nr-axSpA subpopulations at Week 24 | At Week 24
  The ASAS40 response is the relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PtGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
Assessment of SpondyloArthritis International Society 40 % (ASAS40) response criteria in the overall axSpA population, and the AS and nr-axSpA subpopulations at Week 52 | At Week 52
  The ASAS40 response is the relative improvement of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PtGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
Change from Baseline to Week 12 in Bath Ankylosing Spondylitis Functional Index (BASFI) in the overall axSpA population, and the AS and nr-axSpA subpopulations | From Baseline to Week 12
  The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function.
Change from Baseline to Week 24 in Bath Ankylosing Spondylitis Functional Index (BASFI) in the overall axSpA population, and the AS and nr-axSpA subpopulations | From Baseline to Week 24
  The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function.
Change from Baseline to Week 52 in Bath Ankylosing Spondylitis Functional Index (BASFI) in the overall axSpA population, and the AS and nr-axSpA subpopulations | From Baseline to Week 52
  The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function.
Change from Baseline to Week 12 in Patient's Global Assessment of Disease Activity (PtGADA) in the overall axSpA population, and the AS and nr-axSpA subpopulations | From Baseline to Week 12
  Subjects will score their global assessment of their disease activity in response to the question 'how active was your spondylitis on average during the last week?' using a Numeric Rating Scale (NRS) where 0 is 'not active' and 10 is 'very active'.
Change from Baseline to Week 24 in Patient's Global Assessment of Disease Activity (PtGADA) in the overall axSpA population, and the AS and nr-axSpA subpopulations | From Baseline to Week 24
  Subjects will score their global assessment of their disease activity in response to the question 'how active was your spondylitis on average during the last week?' using a Numeric Rating Scale (NRS) where 0 is 'not active' and 10 is 'very active'.
Change from Baseline to Week 52 in Patient's Global Assessment of Disease Activity (PtGADA) in the overall axSpA population, and the AS and nr-axSpA subpopulations | From Baseline to Week 52
  Subjects will score their global assessment of their disease activity in response to the question 'how active was your spondylitis on average during the last week?' using a Numeric Rating Scale (NRS) where 0 is 'not active' and 10 is 'very active'.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (100):
- Belgium (4):
  - 602, Brussels
  - 604, Edegem
  - 601, Genk
  - 603, Heusy
- Germany (43):
  - 53, Altenburg
  - 18, Bayreuth
  - 6, Bayreuth
  - 13, Berlin
  - 14, Berlin
  - 16, Berlin
  - 30, Berlin
  - 7, Berlin
  - 4, Burghausen
  - 25, Chemnitz
  - 50, Cottbus
  - 11, Dresden
  - 8, Düsseldorf
  - 36, Elmshorn
  - 35, Erfurt
  - 19, Freiburg im Breisgau
  - 41, Goslar
  - 26, Greifswald
  - 32, Halle
  - 23, Hamburg
  - 47, Hamburg
  - 1, Hanover
  - 44, Hanover
  - 42, Heidelberg
  - 10, Herne
  - 40, Hofheim am Taunus
  - 34, Hoyerswerda
  - 27, Karlsruhe
  - 48, Karlstadt am Main
  - 49, Karlstadt am Main
  - 21, Leipzig
  - 38, Leipzig
  - 9, Magdeburg
  - 29, Marktredwitz
  - 31, München
  - 43, München
  - 2, Naunhof
  - 20, Planegg
  - 24, Potsdam
  - 15, Püttlingen
  - 28, Saarbrücken
  - 51, Wuppertal
  - 39, Zwickau
- Greece (11):
  - 202, Athens
  - 210, Athens
  - 211, Athens
  - 212, Athens
  - 207, Larissa
  - 208, Marousi
  - 201, Pátrai
  - 203, Thessaloniki
  - 204, Thessaloniki
  - 205, Thessaloniki
  - 206, Thessaloniki
- Italy (6):
  - 504, Florence
  - 501, Palermo
  - 502, Potenza
  - 505, Roma
  - 500, Siena
  - 503, Verona
- Spain (14):
  - 116, Barcelona
  - 114, Bilbao
  - 122, Cartagena
  - 108, Córdoba
  - 118, Donostia / San Sebastian
  - 120, Granada
  - 107, León
  - 123, Lorca
  - 101, Mérida
  - 119, Murcia
  - 117, Salamanca
  - 121, Sant Joan Despí
  - 112, Tarragona
  - 115, Terrassa
- United Kingdom (22):
  - 416, Barnsley
  - 405, Basingstoke
  - 401, Bath
  - 423, Bolton
  - 421, Christchurch
  - 403, Hull
  - 420, Leeds
  - 415, Leicester
  - 409, Liverpool
  - 422, Llandudno
  - 411, Luton
  - 414, Manchester
  - 406, Middlesbrough
  - 424, North Shields
  - 413, Norwich
  - 410, Preston
  - 412, Southampton
  - 419, Stevenage
  - 418, Sunderland
  - 408, Torquay
  - 407, Truro
  - 425, Wigan